CLINICAL TRIAL: NCT03866096
Title: Neuromuscular Training and Strengthening CORE Front of a Neuromuscular Training on Improvement of Knee Stability, Balance and Power in the Vertical Jump in Volleyball Amateur Players. A Randomized Clinical Trial
Brief Title: Neuromuscular Training and Strengthening CORE in Volleyball Amateur Players 18 to 25 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ENCORE
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Stability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Each session will last 20 minutes, taking place during 2 days a week, in a period of 6 weeks. The intervention will be made prior to the training session. The subjects of the experimental group will receive an intervention through neuromuscular training and a CORE strengthening program
  Interventions: Other: Experimental
- Control (Active Comparator): Each session will last 20 minutes, taking place during 2 days a week, in a period of 6 weeks. The intervention will be made prior to the training session. The subjects of the experimental group will receive an intervention through neuromuscular training.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The player will perform exercises of balance, stability, and strengthening of the abdomen, back and gluteus. All these exercises will be carried out in first instance on flat surfaces and later on unstable surfaces to increase the difficulty of it. The training will be done in different levels of difficulty, once the participant managed to master the initial level, advance to the next level to complete the three levels of difficulty during the 6 weeks of training. There will be 3 repetitions of each exercise with a duration of one minute and breaks of 30 seconds between each repetition and 2 minutes of rest between exercises. The duration of the intervention of the experimental group will last 20 minutes
  Other Names: Neuromuscular training and strengthening of CORE
  Arms: Experimental
Other: Control — Neuromuscular training will be applied through balance and stability exercises on both flat and unstable surfaces. There will be 3 repetitions of each exercise with a duration of one minute and breaks of 30 seconds between each repetition and 2 minutes of rest between exercises. The duration of each session of the control group is 10 minutes.
  Other Names: Neuromuscular training
  Arms: Control

SUMMARY:
Introduction. The most popular injuries in volleyball are the ones who occur in knee joints, due the jumps and landings that happen through the game. For this reason there is a high index of loss of stability because of the dynamic valgus during the landing, a loss of balance and a decrease of power during the jumps.

Objective. Evaluate the effectiveness of neuromuscular training in combination with strengthening of CORE in the improvement of knee joint stability, balance and power in vertical jump in volleyball players from 18 to 25 years old.

Study design. Randomized, multicenter, single-blind clinical study with follow-up period.

Methods. The study will be realized with an initial sample of 30 players, which in a random way, will be divided into two groups: experimental and control. It will be realized an initial evaluation where sociodemographic, anthropometric and clinical measures will be taken, and the study variables: knee joint stability (single leg squat test), balance (star excursion balance test) and vertical jump (sargent jump test). The intervention will last six weeks, with two sessions per week of approximately twenty minutes each.

Expected results. The investigators expected to observe improvement in the stability in the knee joint, balance and power in the vertical jump in 18-25 years volleyball players that have received a neuromuscular training with strengthening of CORE.

ELIGIBILITY:
Inclusion Criteria:

* Volleyball players
* Female
* From 18 to 25 years
* With more than one year of sports practice
* Currently participate in amateur industry competitions

Exclusion Criteria:

* Present a medical diagnosis of musculoskeletal injury at the time of beginning the study
* Receive a physiotherapy treatment unrelated to the study
* Have suffered neurological pathology in the last 6 months
* Have some type of auditory or vestibular disorder
* Not signed the informed consent.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline the balance after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Through the Star Excursion Balance test the balance will be assessed, observing the distance (in centimeters) that the subject manages to reach with the unsupported foot. During the test, the player will be placed in standing position performing a monopodal support, asking her to direct the leg that is not supported in the directions: anterior, posterolateral and posteromedial previously drawn on the floor with tape. The evaluator will mark the maximum distance achieved, without moving the support foot and without touching the ground with the reach foot, the subject should not fail when returning the reach foot to the starting position. The greater distance (cm) the better balance. The best of the three attempts made will be taken as a valid measure.

SECONDARY OUTCOMES:
Change from baseline vertical jump power after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Through the Sargent Jump test the vertical jump power will be evaluated, measuring the maximum height (in centimeters) reached during the vertical jump. To perform the test, a tape measure attached to a wall will be placed to measure the height reached. Giving a chalk to the subject so that, from the standing position, lateral to the belt, and with the right arm extended on the head, mark the place where the tips of your fingers reach without lifting the heels of the ground. Once the mark is made, you will be asked to perform the vertical jump, bending the knees, with the left arm attached to the body and the right arm extended over the head. Once in the air, the subject must mark the maximum height obtained on the measuring tape with his fingers. The height of the jump is the difference between the two marks in the tape measure, taking as final value the best of the three jumps, leaving between jump and jump a break of 45 seconds
Change from baseline joint stability of the knee after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Through the Single Leg Squat test the joint stability of the knee will be evaluated, asking the subject to, barefoot, place his hands on the hip, and perform a unipodal squat up to 90 degrees. The participants will perform the test 3 times in a row with each leg. The evaluator will observe any abnormal response that occurs during the performance of the test (shake arms, Trendelenburg sign or valgus or varus support knee collapse). The result will be positive if the participant gets more than two thirds of the abnormal responses in each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided